CLINICAL TRIAL: NCT07109440
Title: The Role of FAPI PET/CT in Exploring the Microenvironment of Colorectal Cancer Liver Metastases: Non-randomized Phase II Molecular Imaging Study
Brief Title: The Role of the Imaging FAPI PET/CT in Exploring the Microenvironment of Colorectal Cancer Liver Metastases
Acronym: FOAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IJB-NM-FOAM
Record Dates: First submitted 2025-07-15; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Liver Metastases From Colorectal Cancer
Keywords: liver metastases from colorectal cancer; FAPI PET/CT; HGP; CAF

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient with liver metastasis from colorectal cancer (Other)
  Interventions: Diagnostic Test: FAPI PET/CT

INTERVENTIONS:
Diagnostic Test: FAPI PET/CT — Patient will undergo FAPI PET/CT Prior to surgery

SUMMARY:
FAPI PET/CT molecular imaging represents a cutting-edge advancement in oncological imaging, particularly for the preoperative assessment of colorectal liver metastases (CRLM). Fibroblast activation protein inhibitors (FAPIs), which are the focus of this imaging modality, selectively target cancer-associated fibroblasts, a critical component of the tumor microenvironment. FAPI PET/CT could be useful in the detection of HGP (Histological Growth Pattern) and in the changes during neoadjuvant chemotherapy prior to surgery

DETAILED DESCRIPTION:
The tumor microenvironment (TME) plays an important role in tumor development and therapeutic response. The understanding of the TME components, especially cancer-associated fibroblasts (CAFs) remains limited. CAFs are among the most abundant and versatile components of the tumor stroma and they are implicated in all the hallmarks of cancer. They have a heterogenous phenotype within a single cell. Some CAFs may have immunosuppressive properties. In liver, there are two obvious physiological sources of CAFs: resident portal fibroblasts (PFs) and hepatic stellate cells (HSCs) . A recent study showed that based on the gene expression profile there are three major subsets of CAFs in colorectal primary tumors and in liver metastasis, including secretory CAFs, ECM-remodeling CAFs and contractile CAFs . In patients undergoing resection of colorectal liver metastasis (CRLMs) the histological growth patterns (HGP) reflect tumor biology and local infiltrating behavior . The HGPs of liver metastases reflect the ways in which cancer cells interact with the surrounding liver. The transition from one HGP to another could occur in patients with CRLM following systemic treatment .

FAPI PET/CT molecular imaging represents a cutting-edge advancement in oncological imaging, particularly for the preoperative assessment of colorectal liver metastases (CRLM). Fibroblast activation protein inhibitors (FAPIs), which are the focus of this imaging modality, selectively target cancer-associated fibroblasts, a critical component of the tumor microenvironment. FAPI PET/CT could be useful in the detection of HGP and in the changes during neoadjuvant chemotherapy prior to surgery

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years.
* Liver metastasis on standard imaging for the initial assessment (MRI, FDG PET/CT)
* Naïve for treatment or after neoadjuvant chemotherapy
* Scheduled for liver metastasis resection
* ECOG Performance status ≤2.
* Signed written informed consent

Exclusion Criteria:

* Non-resectable liver metastases
* Pregnant and lactating women
* Subjects with another significant medical condition which, in the investigator's opinion, may interfere with the completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The quantification of IHC staining for FAP-expressing CAFs measured in patient-derived tissue specimens | from the enrollement to the surgery date, approximately 3 to 4 weeks
The quantification of FAP expression on FAPI PET/CT (SUVmax, SUVmean, MTV [metabolically active tumor volume], FAPI-TV [FAPI positive tumour load]) | From enrollment to surgery date, approximately 3 to 4 weeks
correlation between the value of FAPI PET/CT and the percent encapsulated, and the HGP scores (desmoplastic, replacement, pushing) of the liver metastasis | from the enrollment to the anapathological analysis date,approximately 4 to 5 weeks

SECONDARY OUTCOMES:
Correlation between FAPI PET/CT and FDG PET/CT parameters: (SUV max, SUVmean, metabolical volume) | from enrollment to the surgery date, approximately 3 to 4 weeks
Correlation between FAPI metabolical volume and MRI tumor volume | from enrollment to the surgery date, approximately 3 to 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jules Bordet, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided